CLINICAL TRIAL: NCT03530202
Title: The Effect of High-velocity Resistance Training (HVRT) and Creatine Supplementation in Healthy Aging Males
Brief Title: Effects of High-velocity Resistance Training and Creatine Supplementation in Healthy Aging Males
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Regina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: URegina
Record Dates: First submitted 2018-04-19; First posted 2018-05-21 (Actual); Last update posted 2018-05-21 (Actual); Status verified 2018-05

CONDITIONS: Sarcopenia
Keywords: muscle thickness; strength; power; functionality
MeSH Terms: conditions — Sarcopenia | interventions — Creatine

STUDY DESIGN:
Intervention Model Description: The study will be a double-blind, repeated measures design. Participants will be randomized on a 1:1 basis to one of two groups: high-velocity resistance training and creatine or high-velocity resistance training and placebo.
Who Masked: Participant, Investigator
Masking Description: A research assistant who is not involved in the study in any other way will be responsible for randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HVRT + Creatine Monohydrate (Experimental): Participants will perform 8-weeks of high-velocity resistance training, defined as performing the concentric phase of a lift as fast as possible and taking two seconds to perform the eccentric phase of the lift, on six exercises (bilateral legpress, leg extension, leg curl, chest press, triceps extension, and biceps curl) and consume creatine monohydrate powder. The load will be 80% of the participants one-repetition max (1RM; the maximum weight that can be successfully lifted one time with proper form).
  Interventions: Drug: Creatine monohydrate
- HVRT + Maltodextrin Powder (Placebo Comparator): Participants will perform 8-weeks of high-velocity resistance training, defined as performing the concentric phase of a lift as fast as possible and taking two seconds to perform the eccentric phase of the lift, on six exercises (bilateral legpress, leg extension, leg curl, chest press, triceps extension, and biceps curl) and consume maltodexterin powder. The load will be 80% of the participants one-repetition max (1RM; the maximum weight that can be successfully lifted one time with proper form).
  Interventions: Drug: Maltodextrin Powder

INTERVENTIONS:
Drug: Creatine monohydrate — Participants will consume creatine monohydrate powder (Creapure, AlzChem AG, Trostberg, Germany) every day for 8 weeks. On training days participants will consume supplement immediately after each training session (~ 5 minutes) mixed in water as post-exercise creatine ingestion enhances its uptake into muscle and promotes increased muscle mass. On non-training days, supplements will be consumed at the participant's leisure.
  Other Names: Creapure, AlzChem AG, Trostberg, Germany
  Arms: HVRT + Creatine Monohydrate
Drug: Maltodextrin Powder — Participants will consume Maltodextrin Powder (Globe Plus 10 DE Maltodextrin Powder, Univar Canada) every day for 8 weeks. On training days participants will consume supplement immediately after each training session (~ 5 minutes) mixed in water. On non-training days, supplements will be consumed at the participant's leisure.
  Other Names: Globe Plus 10 DE Maltodextrin, Univar, Canada
  Arms: HVRT + Maltodextrin Powder

SUMMARY:
The age-related loss of skeletal muscle mass (i.e. sarcopenia)and muscle performance (i.e. strength and power), decreases functionality and the ability to perform activities of daily living. Therefore, lifestyle interventions which may improve aging muscle health are important (i.e. resistance training and creatine supplementation). High-velocity resistance training (HVRT) has been shown to increase muscle mass and muscle performance in aging adults. Creatine (CR), a compound naturally found in red meat and seafood, has also been shown to increase muscle mass and muscle performance in aging adults. No study has examined the combined effects of HVRT and CR supplementation in aging adults. This study may determine whether this lifestyle intervention is effective to combat sarcopenia.

DETAILED DESCRIPTION:
Purpose and hypothesis: The purpose of this thesis is to compare the effects of HVRT and CR supplementation to HVRT and placebo in healthy aging males. It is hypothesized that HVRT and CR supplementation will increase muscle mass, strength, power and tasks of functionality compared to HVRT and placebo.

Participants: An a priori power analysis (G*Power v. 3.1.5.1) indicated that 34 participants are required. This is based on a moderate effect size (Cohen's d = 0.25), an alpha level of .05, a ß-value of 0.8 for a repeated measures, within-between analysis of variance (ANOVA) design. Males (≥ 50 years) who are not engaged in resistance training for ≥ 6 weeks prior to the start of the study will be recruited. Participants will be informed of the risks and purposes of the study before written consent is obtained. The study will be approved by the Research Ethics Board at the University of Regina.

Methods and Research Design: The study will be a double-blind, repeated measures design. Participants will be randomized on a 1:1 basis to one of two groups: HVRT and CR or HVRT and placebo. The CR dosage will be 0.1g/kg/day as this dosage is effective for increasing muscle mass in aging males without resulting in adverse effects. On training days, participants will consume their supplement immediately after each training session mixed in water, juice or milk as post-exercise CR ingestion enhances its uptake into muscle and promotes increased muscle mass.

High-velocity Resistance Training Program: Participants will perform 3 sets of repetitions at 80% baseline 1-repetition maximum (1-RM) for the leg press, leg extension, leg curl, chest press, biceps curl, and triceps extension 2 times per week, for 8 weeks. Participants will perform the concentric phase of each muscle contraction as quickly as possible and will take 2 seconds to perform the eccentric phase.

Primary Dependent Variables

1. Muscle thickness: Muscle thickness will be assessed by B-mode ultrasound (LOGIQ e, GE Medical Systems) on knee flexors, knee extensors, elbow flexors, and elbow extensors in the Aging Muscle and Bone Health Laboratory, University of Regina.
2. Muscle strength: Leg press and chest press strength will be assessed using a 1-RM testing procedure in the Aging Muscle and Bone Health Laboratory, University of Regina.
3. Muscle power: Torque (Nm) and power (watts) will be measured for the knee flexors and extensors using an isokinetic dynamometer (Biodex System 3, Biodex Medical Systems Inc.).
4. Functionality tests: Dynamic balance will be measured as the time taken to perform backwards tandem walking over a distance of 6m on a 10cm-wide board that is raised about 4cm off the ground. Walking speed will be assessed by the time needed to walk an 80 m course.

Statistical Analyses: A 2 (group: CR vs. placebo) x 2 (time: pre- vs. post-training) repeated measures ANOVA will be used to determine differences between groups over time for the dependent variables. A one-factor ANOVA will be used to assess baseline characteristics and total training volume between groups. Significance will be set at an alpha level of 0.05 and all results will be expressed as means ± standard deviation. The magnitude of the difference between significant means will be determined by eta squared (η2). Statistical analyses will be performed using IBM SPSS Statistics, v. 24.

ELIGIBILITY:
Inclusion Criteria:

* Males (≥ 50 years) who are not engaged in supervised resistance training for ≥ 6 weeks prior to the start of the study will be recruited to participate.

Exclusion Criteria:

* Participants will be excluded if they have taken medications that affect muscle biology or creatine monohydrate ≤ 12 weeks prior to the start of the study
* If they have a history of fragility fractures; diseases that are known to affect muscle biology (i.e. corticoids)
* If they suffer from severe osteoarthritis
* If they are currently participating in moderate-vigorous resistance training (≥ 3 times per week)
* If they are vegetarian
* If they are planning to travel during the study period for greater than 2 weeks duration at a time.
* Participants with kidney or liver abnormalities will be excluded.

Min Age: 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — The response to creatine supplementation is inconsistent between males and females. Females may not experience the same gains in muscle mass and strength following creatine supplementation and resistance training compared to males. Although speculative, females may have higher initial intramuscular creatine stores than males which make them less responsive to supplementation. Furthermore, creatine appears to have no effect on muscle protein kinetics in females. Therefore, for the purpose of this study, only healthy aging males will be recruited.
Enrollment: 40 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-07-31 (Estimated); Study Completion 2018-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in muscle thickness | Baseline and again once intervention is completed (8 weeks)
  Muscle thickness (right side) of the elbow flexors, elbow extensors, knee flexors, and knee extensors will be measured using B-Mode ultrasound (LOGIQ e, GE Medical Systems).

SECONDARY OUTCOMES:
Change in muscle strength | Baseline and again once intervention is completed (8 weeks)
  Leg press and chest press strength will be assessed using a 1-repetition maximum (1-RM) standard testing procedure in the Aging Muscle and Bone Health Laboratory, University of Regina.
Change in peak torque (Nm) | Baseline and again once intervention is completed (8 weeks)
  Peak torque (Nm) will be measured for the knee flexors and extensors using an isokinetic dynamometer (Biodex System 3, Biodex Medical Systems Inc.).
Change peak muscle power (watts) | Baseline and again once intervention is completed (8 weeks)
  Peak muscle power (watts) will be measured for the knee flexors and extensors using an isokinetic dynamometer (Biodex System 3, Biodex Medical Systems Inc.).
Change in dynamic balance | Baseline and again once intervention is completed (8 weeks)
  Dynamic balance will be measured as the time taken to perform backwards tandem walking (i.e. toe to heel) over a distance of 6m on a 10cm-wide board that is raised about 4cm off the ground.
Walking speed | Baseline and again once intervention is completed (8 weeks)
  Walking speed will be assessed by the time needed to walk an 80 m course at a fast pace.

CONTACTS AND LOCATIONS:
Overall Officials: Darren G Candow, PhD, Principal Investigator — Professor, Associate Dean of Graduate Studies
Locations (1):
- University of Regina, Regina, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Background] Candow DG, Little JP, Chilibeck PD, Abeysekara S, Zello GA, Kazachkov M, Cornish SM, Yu PH. Low-dose creatine combined with protein during resistance training in older men. Med Sci Sports Exerc. 2008 Sep;40(9):1645-52. doi: 10.1249/MSS.0b013e318176b310. PMID 18685526
- [Background] Chilibeck PD, Stride D, Farthing JP, Burke DG. Effect of creatine ingestion after exercise on muscle thickness in males and females. Med Sci Sports Exerc. 2004 Oct;36(10):1781-8. doi: 10.1249/01.mss.0000142301.70419.c6. PMID 15595301
- [Background] Harris RC, Soderlund K, Hultman E. Elevation of creatine in resting and exercised muscle of normal subjects by creatine supplementation. Clin Sci (Lond). 1992 Sep;83(3):367-74. doi: 10.1042/cs0830367. PMID 1327657
- [Background] Nogueira W, Gentil P, Mello SN, Oliveira RJ, Bezerra AJ, Bottaro M. Effects of power training on muscle thickness of older men. Int J Sports Med. 2009 Mar;30(3):200-4. doi: 10.1055/s-0028-1104584. Epub 2009 Feb 6. PMID 19199198